CLINICAL TRIAL: NCT00256269
Title: A Phase II Study of Weekly Oxaliplatin and Irinotecan in the Treatment of Recurrent or Metastatic Esophageal Carcinoma and Carcinoma of the Gastroesophageal (GE) Junction
Brief Title: Oxaliplatin and Irinotecan in Recurrent or Metastatic Esophageal and Gastroesophageal (GE) Junction Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated by funding entity
Sponsor: University of California, Irvine (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Sai-Hong Ignatius Ou, HS Associate Clinical Professor, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCI 04-09; 2004-3849 (Other: University of California, Irvine)
Record Dates: First submitted 2005-11-17; First posted 2005-11-21 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Esophageal Cancer; Gastroesophageal Cancer
Keywords: Esophageal Cancer; Gastroesophageal junction cancer; Oxaliplatin; Irinotecan
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Oxaliplatin; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Oxaliplatin plus Irinotecan (Experimental): Drug: Oxaliplatin-40 mg/m2 IV over 60 minutes Every 21 days. Drug: Irinotecan-60 mg/m2 IV over 60 minutes, immediately following oxaliplatin Every 21 days.
  Interventions: Drug: Oxaliplatin; Drug: Irinotecan

INTERVENTIONS:
Drug: Oxaliplatin — 40 mg/m2 IV over 60 minutes Every 21 days
Drug: Irinotecan — 60 mg/m2 IV over 60 minutes, immediately following oxaliplatin Every 21 days

SUMMARY:
The combination of cisplatin and irinotecan has significant anti-tumor activity in esophageal cancer. Oxaliplatin has been shown to have activity in combination with 5-Fluorouracil (5FU) and radiation in treatment of locally advanced esophageal cancer. Oxaliplatin also has better side effects profile than cisplatin and may be able to overcome tumors that have developed cisplatin resistance. The standard treatment of locally advanced esophageal cancer has been cisplatin, 5FU and radiation followed by possible esophagectomy. However, a large portion of these patients will relapse and the tumor may develop resistance to cisplatin and/or the cumulative toxicity from previous treatment forbids the use of cisplatin again. Weekly combination of oxaliplatin and irinotecan has been shown to be active and well tolerated in elderly population with refractory colorectal cancer. Therefore, we propose this phase II trial of a weekly oxaliplatin and irinotecan to test the effectiveness and the tolerability of this regimen in metastatic and/or recurrent esophageal cancer.

DETAILED DESCRIPTION:
Esophageal cancer represents the seventh cause of cancer death in American men, and more than 90% of patients diagnosed with esophageal cancer will ultimately die of their disease. In the United States, 13,900 new cases of esophageal cancer and 13,000 deaths from esophageal cancer are anticipated in 2003 (Jemal et al, 2003). The lifetime risk of esophageal cancer is 0.8% for men and 0.3% for women (Ries et al, 2002). The risk increases with age, with a mean age at diagnosis of 67 years (Ries et al, 2002; Daly et al, 2000). Adenocarcinoma of the esophagus or gastroesophageal junction, a previously rare disease, is rapidly increasing in incidence in the United States and western countries and now accounts for more than half of newly diagnosed disease (Devesa et al, 1998).

Half of patients diagnosed with esophageal cancer present with overt metastatic disease, and chemotherapy is the mainstay of palliation in this setting. In patients who present initially with locoregional disease, the majority will eventually develop metastatic disease as well, with or without local recurrence of disease. Metastatic esophageal carcinoma is an incurable disease with median survival duration of 4 to 8 months. Combination chemotherapy, most often cisplatin-based, results in partial responses in 25% to 50% of patients with metastatic disease and rare complete responses, including a 35% response rate reported for the commonly used combination of cisplatin and fluorouracil (Ilson et al, 1996). Recent chemotherapy trials indicate an overlap in response rates for metastatic adenocarcinoma and squamous carcinoma carcinoma of the esophagus (Ilson et al, 1997). Responses to chemotherapy are generally short-lived, and toxicity of cisplatin-based chemotherapy, particularly in the palliation of metastatic disease, is often substantial and underscores the need to identify new agents in the treatment of esophageal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have histologically or cytologically confirmed diagnosis of squamous cell carcinoma or adenocarcinoma of the esophagus. Patients with tumors of the gastroesophageal junction were eligible if at least 50% of the tumor involved the esophagus.
* Patients must have locally advanced (i.e. unresectable) or metastatic disease
* All sites of disease must be assessed and designated as measurable or non-measurable disease as documented by CT, MRI, X-ray physical Each of the criteria in the following section must be met in order for a patient to be eligible for registration.
* Patients may have received prior radiotherapy if there has been complete recovery from all radiation-induced toxicities. At least 4 weeks must have been elapsed from the completion of radiation therapy to the time of registration. If lesions within the radiation port are to be used to assess response to therapy, those lesions must have demonstrated clear progression by the criteria outlined in Section 10.2d following completion of radiation therapy.
* Patients must have adequate bone marrow reserve as documented by absolute neutrophil count (ANC) > 1,500 microliters and platelets > 100,000/microliter obtained within 14 days prior to registration.
* Patients must have adequate hepatic as documented by serum bilirubin < 1.5 x the institutional upper limit of normal. Serum transaminase (SGOT or SGPT) must be < 1.5 x the institutional upper limit of normal serum unless the liver is involved with tumor, in which case serum transaminase (SGOT or SGPT) must be < 5 x the institutional limit of normal. These tests must be obtained within 14 days prior to registration.

Patients must have a creatinine < 1.5 x the institutional upper limit of normal or a creatinine clearance of > 30 cc/min calculated using the following formula obtained within 28 days prior to registration.

Calculated Creatinine Clearance = (140-age) X wt (kg) X (0.85 if female) 72 X creatinine (mg/dl)

These tests must have been performed within 28 days prior to registration.

* All patients must be 18 years of age or older
* Patients must have a Zubrod performance of 0-2

Exclusion Criteria:

* Patients must not have received prior chemotherapy for chemotherapy for advanced or metastatic esophageal cancer. Chemotherapy given adjuvantly or as a radiosensitizer is allowed if more than 8 weeks have elapsed since the treatment was completed and they have recovered from any treatment related toxicity.
* Patients must not have a surgical procedure for esophageal cancer within 4 weeks prior to registration. Patients must have completely recovered from all surgery prior to registration.
* Patients with any evidence of active or uncontrolled infection, recent myocardial infection, unstable angina, or life-threatening arrhythmia are not eligible.
* Patients with severe psychiatric disorder are not eligible.
* Patients with known brain metastasis are not eligible. However, brain-imaging studies are not required for eligibility if the patient has no neurological signs or symptoms. If brain-imaging studies are performed, they must be negative for disease.
* No other prior malignancy is allowed except for adequately treated basal cell or squamous cell carcinoma, in situ cervical cancer, or adequately treated Stage I and II cancer from which the patient is in complete remission, or any other malignancy from which the patient has been disease-free for 5 years.
* Patients should not have active infection.
* Patients should not have psychological, familial, sociological, or geographical conditions that do not permit medical follow-up and compliance with study protocol.
* Except for cancer-related abnormalities, patients should not have unstable or pre-existing major medical conditions.
* Patients should not have any immediate life-threatening complications of their malignancies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2005-06 (Actual); Primary Completion 2007-02-07 (Actual); Study Completion 2007-02-07 (Actual)

PRIMARY OUTCOMES:
To assess the overall response rate | 5 years
  To assess the overall response rate (complete and partial response) to a weekly combination of oxaliplatin and irinotecan in patients with unresectable or metastatic esophageal cancer or cancer of the gastro-esophageal (GE) junction.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v3.0 | 5 years
  To assess the frequency and severity of toxicities associated with this treatment
Progression Free Survival | 5 years
  from date of registration to date of first observation of progressive disease (as outlined in 10.2d), death due to any cause or symptomatic deterioration.
Evaluation of Time to Death | 5 years
  Analysis timeline would be from the date of registration to date of death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Sai-Hong Ignatius Ou, MD, Principal Investigator — Chao Family Comprehensive Cancer Center
Locations (1):
- Chao Family Comprehensive Cancer Center, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No